CLINICAL TRIAL: NCT03722589
Title: Randomized Open-Label Trial to Compare the Immunogenicity of Cell Culture-Based and Recombinant Unadjuvanted Quadrivalent Influenza Vaccines to Conventional Egg-Based Unadjuvanted Quadrivalent Influenza Vaccines Among Healthcare Personnel Aged 18-64 Years
Brief Title: Immunogenicity Trial of Egg- Versus Non-Egg-Based Influenza Vaccines Among HCP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Baylor Scott and White Health (Other); Kaiser Permanente (Other); Abt Associates (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7179
Record Dates: First submitted 2018-10-15; First posted 2018-10-29 (Actual); Results first posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluBlok; Influenza Vaccines; fluarix; Fluzone High-Dose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Flublok (Recombinant) (Active Comparator): Flublok® Quadrivalent by Sanofi Pasteur, 45µg of HA per strain
  Interventions: Biological: Flublok
- Flucelvax (Cell-based) (Active Comparator): Flucelvax™ Quadrivalent by Seqirus, Inc., 15µg of HA per strain
  Interventions: Biological: Flucelvax
- Fluarix (Egg-based) (Active Comparator): Fluarix® Quadrivalent by GlaxoSmithKlein, 15µg of HA per strain
  Interventions: Biological: Fluarix
- Fluzone (Egg-based) (Active Comparator): Fluzone® Quadrivalent by Sanofi Pasteur, 15µg of HA per strain
  Interventions: Biological: Fluzone
- Fluzone (Egg-based) High-Dose (Active Comparator): Fluzone® Trivalent High-Dose by Sanofi Pasteur, 60µg of HA per strain
  Interventions: Biological: Fluzone High-Dose

INTERVENTIONS:
Biological: Flublok — 0.5 mL intramuscular dose of Flublok
  Arms: Flublok (Recombinant)
Biological: Flucelvax — 0.5 mL intramuscular dose of Flucelvax
  Arms: Flucelvax (Cell-based)
Biological: Fluarix — 0.5 mL intramuscular dose of Fluarix
  Arms: Fluarix (Egg-based)
Biological: Fluzone — 0.5 mL intramuscular dose of Fluzone
  Arms: Fluzone (Egg-based)
Biological: Fluzone High-Dose — 0.5 mL intramuscular dose of Fluzone
  Arms: Fluzone (Egg-based) High-Dose

SUMMARY:
This randomized, open-label trial will assess humoral and cell-mediated immune responses to cell culture-based and recombinant unadjuvanted quadrivalent influenza vaccines compared to conventional egg-based unadjuvanted quadrivalent standard dose (15µg of HA per strain) influenza vaccines among persons aged 18-64 years. The trial will be conducted at two sites in the United States during two influenza seasons (2018-19 and 2019-20). Stratified enrollment procedures will be used to enroll a mix of participants based on age.

DETAILED DESCRIPTION:
In year 1 of the trial (the 2018-19 Northern Hemisphere influenza season), eligible participants at each site will be randomized 2:2:1:1 to receive a single dose of cell culture-based vaccine (Flucelvax™ Quadrivalent by Seqirus, Inc., 15µg of HA per strain) versus recombinant vaccine (Flublok® Quadrivalent by Sanofi Pasteur, 45µg of HA per strain) versus one of two standard dose egg-based vaccines (Fluzone® Quadrivalent by Sanofi Pasteur, 15µg of HA per strain and Fluarix® Quadrivalent by GlaxoSmithKlein, 15µg of HA per strain) during August-September of 2018. All study vaccines are licensed for use in adults aged >18 years in the United States. Participants will have blood collected just prior to vaccination and at approximately 28 days and 6 months post-vaccination (or at the end of influenza virus circulation as determined by available surveillance data) to evaluate humoral immune responses to vaccination.

In year 1, sites will aim to enroll 864 participants (432 per site) at the start of the 2018-19 season, including up to 200 participants (up to 100 per site) who will contribute additional blood at all study visits to evaluate cell-mediated immune responses to vaccination. Efforts will be made to retain participants enrolled in the first year of the study for both years of the study. Sites will also enroll additional participants at the start of the 2019-20 season to make up for participants who withdraw or are lost to follow-up prior to the start of the 2019-20 season. Both participants and study investigators will be aware of study arm assignments with the exception of laboratory investigators who will be blinded to study arm assignment until testing is completed, as appropriate.

In year 1 , relative efficacy of single doses of study vaccines will be assessed by comparing immunologic responses to vaccination among participants between study arms using Fluzone® Quadrivalent and Fluarix® Quadrivalent as the comparator groups for participants in the Flucelvax™ Quadrivalent or Flublok® Quadrivalent arms. In addition, the effect of frequency of prior vaccination during the preceding five years on immunologic responses to vaccine will be evaluated in subgroup analysis. Both humoral (influenza antibody) and cell-mediated (influenza- specific CD4 and CD8 T cell) immune responses will be evaluated.

In year 2 of the trial, (the 2019-20 Northern Hemisphere influenza season), participants from the first year of the trial who received Flucelvax™ Quadrivalent or Flublok® Quadrivalent will be randomized 1:1 to receive Flucelvax™ Quadrivalent or Flublok® Quadrivalent, and participants who received an egg-based standard-dose vaccine in year one (Fluzone® Quadrivalent or Fluarix Quadrivalent) will be randomized 1:1:1 to receive Flucelvax™ Quadrivalent , Flublok® Quadrivalent , or Fluzone® Quadrivalent. In addition, both sites will enroll additional participants in year 2 to achieve a total of 150 participants per site (including participants who continue from year one plus additional newly enrolled participants) who received egg-based standard dose influenza vaccine during the 2018-2019 influenza season and who will be randomized 1:1:1 to receive Flucelvax™ Quadrivalent, Flublok® Quadrivalent, or Fluzone® Quadrivalent in year two. The Kaiser Permanente Northwest site site will also enroll up to 80 new participants for a non-randomized study arm that will receive Fluzone® High-Dose. All study vaccines except Fluzone High-Dose are licensed for use in adults aged >=18 years in the United States. Fluzone High-Dose is licensed for use in adults aged >=64 years in the United States and will be used off-label in this trial. Participants will have blood collected just prior to vaccination and at approximately 28 days post-vaccination (or at the end of influenza virus circulation as determined by available surveillance data) to evaluate humoral immune responses to vaccination. Additional blood will be collected from a subset of participants pre-vaccination and at approximately 7 and 28 days post-vaccination to evaluate cell-mediated immune responses to vaccination.

In year 2, sites will aim to retain from year 1 or newly enroll 750 participants.

Deaths and/or adverse events were not monitored/assessed in any arms for any flu seasons

ELIGIBILITY:
Inclusion Criteria:

* Healthcare personnel (HCP) who have direct contact with patients, including dentists and other dental health personnel
* Enrolled in Scott & White Healthcare or Kaiser Permanente health network for at least one month
* Aged 18-64 years for newly enrolled participants
* Aged 18-65 years for participants who were originally enrolled in year one of the study and return for year 2
* Available and willing to participate in study follow-up through the end of the 2019-2020 influenza season (i.e. at least approximately 18 months if enrolled during season 1 or 6 months if enrolled during season 2)
* Received an egg-based standard dose influenza vaccine during the 2018-2019 influenza season (for participants enrolled for the first-time during year two)

Exclusion Criteria:

* Already received an influenza vaccine during the current influenza season
* Previous hypersensitivity reaction to the study vaccines as reported by the subject
* Received any vaccine in the 4 weeks prior to the first study visit or plans to receive a vaccine (other than influenza vaccine provided through the study protocol) in the 4 weeks following the first study visit
* Currently participating in a study that involves an experimental agent (vaccine, drug, biologic, device, blood product, or medication), or has received an experimental agent within 1 month prior to enrollment in this study, or expects to receive an experimental agent during participation in this study
* Any condition that the principle investigator (PI) believes may interfere with successful completion of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 944 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fatimah Dawood, MD, Principal Investigator — Centers for Disease Control and Prevention; Brendan Flannery, PhD, Principal Investigator — Centers for Disease Control and Prevention
Locations (2):
- United States (2):
  - Kaiser Permanente Northwest, Portland, Oregon
  - Baylor Scott and White Health, Temple, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available to contractor and site research staff. This data can be made available to other researchers upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Study period

REFERENCES:
- [Derived] Liu F, Gross FL, Joshi S, Gaglani M, Naleway AL, Murthy K, Groom HC, Wesley MG, Edwards LJ, Grant L, Kim SS, Sambhara S, Gangappa S, Tumpey T, Thompson MG, Fry AM, Flannery B, Dawood FS, Levine MZ. Redirecting antibody responses from egg-adapted epitopes following repeat vaccination with recombinant or cell culture-based versus egg-based influenza vaccines. Nat Commun. 2024 Jan 4;15(1):254. doi: 10.1038/s41467-023-44551-x. PMID 38177116
- [Derived] Gaglani M, Kim SS, Naleway AL, Levine MZ, Edwards L, Murthy K, Dunnigan K, Zunie T, Groom H, Ball S, Jeddy Z, Hunt D, Wesley MG, Sambhara S, Gangappa S, Grant L, Cao W, Gross FL, Mishina M, Fry AM, Thompson MG, Dawood FS, Flannery B. Effect of Repeat Vaccination on Immunogenicity of Quadrivalent Cell-Culture and Recombinant Influenza Vaccines Among Healthcare Personnel Aged 18-64 Years: A Randomized, Open-Label Trial. Clin Infect Dis. 2023 Feb 8;76(3):e1168-e1176. doi: 10.1093/cid/ciac683. PMID 36031405
- [Derived] Dawood FS, Naleway AL, Flannery B, Levine MZ, Murthy K, Sambhara S, Gangappa S, Edwards L, Ball S, Grant L, Belongia E, Bounds K, Cao W, Gross FL, Groom H, Fry AM, Rentz Hunt D, Jeddy Z, Mishina M, Kim SS, Wesley MG, Spencer S, Thompson MG, Gaglani M. Comparison of the Immunogenicity of Cell Culture-Based and Recombinant Quadrivalent Influenza Vaccines to Conventional Egg-Based Quadrivalent Influenza Vaccines Among Healthcare Personnel Aged 18-64 Years: A Randomized Open-Label Trial. Clin Infect Dis. 2021 Dec 6;73(11):1973-1981. doi: 10.1093/cid/ciab566. PMID 34245243

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During year 1, participants were randomized to 1 of 4 vaccine assignments as shown. During year 2, some participants from year 1 were retained (n=546) and additional participants (n=217) were enrolled. During year 2, retained participants from year 1 were rerandomized to vaccine groups. Participants completed consent at year 1 start and again at year 2 start, so the number of enrolled participants at year 2 start is not the cumulative sum of participants enrolled at year 1 and year 2 start.
Period: Year 1 (2018-19)
Arm/Group | Flublok (Recombinant) | Flucelvax (Cell-based) | Fluarix (Egg-based) | Fluzone (Egg-based) | Fluzone (Egg-based) High-Dose
Started | 202 | 283 | 120 | 122 | 0
Completed | 195 | 279 | 97 | 86 | 0
Not Completed | 7 | 4 | 23 | 36 | 0
Period: Year 2 (2019-20)
Arm/Group | Flublok (Recombinant) | Flucelvax (Cell-based) | Fluarix (Egg-based) | Fluzone (Egg-based) | Fluzone (Egg-based) High-Dose
Started | 292 (Additional participants were enrolled between year 1 and year 2 and some participants from year 1 did not consent to continued enrollment in year 2; therefore the number of participants completing year 1 is not equal to the number of participants starting year 2.) | 287 (Additional participants were enrolled between year 1 and year 2 and some participants from year 1 did not consent to continued enrollment in year 2; therefore the number of participants completing year 1 is not equal to the number of participants starting year 2.) | 0 (Additional participants were enrolled between year 1 and year 2 and some participants from year 1 did not consent to continued enrollment in year 2; therefore the number of participants completing year 1 is not equal to the number of participants starting year 2.) | 105 (Additional participants were enrolled between year 1 and year 2 and some participants from year 1 did not consent to continued enrollment in year 2; therefore the number of participants completing year 1 is not equal to the number of participants starting year 2.) | 79 (Additional participants were enrolled between year 1 and year 2 and some participants from year 1 did not consent to continued enrollment in year 2; therefore the number of participants completing year 1 is not equal to the number of participants starting year 2.)
Completed | 285 | 281 | 0 | 103 | 79
Not Completed | 7 | 6 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for Year 1 participants. There were no Fluzone High-Dose participants enrolled in year 1.
Groups:
- Fluzone High Dose - Year 2: Fluzone High Dose by Sanofi Pasteur, 45µg of HA per strain
  Fluzone High Dose: 0.5 mL intramuscular dose of Fluzone
- Total: Total of all reporting groups
Arm/Group | Flublok (Recombinant) | Flucelvax (Cell-based) | Fluarix (Egg-based) | Fluzone (Egg-based) | Fluzone High Dose - Year 2 | Total
Number analyzed (Participants) | 202 | 283 | 120 | 122 | 79 | 806
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 202 | 283 | 120 | 122 | 79 | 806
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 232 | 103 | 107 | 53 | 652
  Male | 45 | 51 | 17 | 15 | 26 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 37 | 19 | 13 | 4 | 110
  Not Hispanic or Latino | 165 | 246 | 101 | 109 | 75 | 696
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 202 | 283 | 120 | 122 | 79 | 806

OUTCOME MEASURES:

1. Primary Outcome: Microneutralization (MN) Assay Response to Cell-grown Influenza A/H3N2 - Seroconversion Rate (SCR)
Description: MN responses to the cell-grown influenza A/H3N2 vaccine reference viruses for each study season at approximately 28 days post-vaccination, including by assessing SCR in the various vaccine arms defined as the proportion of participants with paired samples that achieved ≥ 4 fold rises comparing post- versus pre-vaccination titers, and post vaccination titers ≥ 40
Time Frame: 28 days post-vaccination during year 1
Population: For the primary analysis, the Fluarix and Fluzone arms were combined as prespecified in the study protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Fluarix (Egg-based)/Fluzone (Egg-based): Fluarix® Quadrivalent by GlaxoSmithKlein, 15µg of HA per strain
  Fluarix: 0.5 mL intramuscular dose of Fluarix
Arm/Group | Flublok (Recombinant) | Flucelvax (Cell-based) | Fluarix (Egg-based)/Fluzone (Egg-based)
Number analyzed (Participants) | 202 | 283 | 242
Participants | 112 | 48 | 29

2. Primary Outcome: Microneutralization (MN) Assay Response to Cell-grown Influenza A/H3N2 - Seroconversion Rate (SCR)
Description: as for outcome 1
Time Frame: 28 days post-vaccination during year 2
Population: For the primary analysis, the Fluarix and Fluzone arms were combined as prespecified in the study protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Fluzone High Dose: Fluzone® High Dose by Sanofi Pasteur, 45µg of HA per strain
  Fluzone High Dose: 0.5 mL intramuscular dose of Fluzone
Arm/Group | Flublok (Recombinant) | Flucelvax (Cell-based) | Fluzone (Egg-based) | Fluzone High Dose
Number analyzed (Participants) | 103 | 106 | 102 | 79
Participants | 103 | 106 | 102 | 79

ADVERSE EVENTS:
Time Frame: Solicited adverse event information was not collected in this trial.
Description: Deaths and/or adverse events were not monitored/assessed in any arm of this study.
Arm/Group | Flublok (Recombinant) | Flucelvax (Cell-based) | Fluarix (Egg-based) | Fluzone (Egg-based)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Original Protocol and Statistical Analysis Plan, Year 1 (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/89/NCT03722589/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Year 2 Protocol Amendment (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT03722589/Prot_SAP_003.pdf